CLINICAL TRIAL: NCT06601257
Title: An Open-Label, Single-Dose, Pharmacokinetic Study of Vancomycin Dosed by Weight or Kidney Function in Adults With Obesity
Brief Title: Vancomycin Dose Optimization in Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Manjunath Prakash Pai, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00256444; 75F40122C00147 (Other Grant/Funding Number: Health and Human Services, Department of-Food and Drug Administration)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pharmacokinetics and Pharmacodynamics
Keywords: obesity; pharmacokinetics; vancomycin; antibiotics; body composition; kidney function; renal
MeSH Terms: conditions — Obesity | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Weight-stratified dosing as the current standard of care
  Interventions: Drug: Vancomycin (IV)
- Test (Experimental): Kidney function stratified dosing
  Interventions: Drug: Vancomycin (IV)

INTERVENTIONS:
Drug: Vancomycin (IV) — Vancomycin weight-based or kidney function-based dosing

SUMMARY:
The goal of this clinical trial is to learn how to optimize vancomycin dosing in obese adults based on weight and kidney function. It will also assess the safety of different vancomycin dosing strategies. The main questions it aims to answer are:

Does dosing vancomycin based on kidney function provide better drug exposure than dosing based on weight? What medical or safety issues arise when vancomycin is dosed according to weight versus kidney function? Participants will be randomized into two groups. One group will receive vancomycin doses based on their weight, while the other will receive doses based on their kidney function.

Participants will:

Receive a single dose of vancomycin based on either their weight or kidney function after pretreatment with antihistamines Provide blood and urine samples at specific times for pharmacokinetic analysis Undergo body composition measurements using DEXA scans and other methods Visit the clinic for physical exams, medical history, and laboratory tests

DETAILED DESCRIPTION:
This prospective, dosing group-randomized, single-dose pharmacokinetic study aims to evaluate vancomycin dosing in healthy obese participants across three BMI and two kidney function categories. Twenty-four participants will be enrolled, stratified by BMI (30-34.9 kg/m², 35-39.9 kg/m², ≥40 kg/m²) and creatinine clearance using dosing weight (CLcr_dw 60-119 mL/min or ≥120 mL/min). Twenty-four participants will be randomized (1:1) into a standard of care vancomycin group (Control) or a kidney function based group (Test). The study will include physical exams, medical history, and laboratory evaluations. Vancomycin doses will be administered based on weight or kidney function after pretreatment with antihistamines. Pharmacokinetic data will be collected through blood and urine samples at specific time points. Body composition measurements will be performed using DEXA and through anthropometric methods. Serum cystatin C concentrations will also be measured. Data analysis will include fitting vancomycin concentration-time data using a 2-compartment linear model to estimate area under the curve (AUC). Group comparisons for AUC target attainment (400-600 h*mg/L) will be performed using Fisher's Exact Test. Additionally, the study will test if the investigators can reduce the standard two-sample method for AUC estimation to a single sample. Different models of estimated glomerular filtration rate (eGFR) will be compared as predictors of vancomycin clearance (CL). This study will provide insights into optimizing vancomycin dosing in obese individuals with varying kidney function, potentially improving therapeutic drug monitoring strategies.

ELIGIBILITY:
Inclusion Criteria:

1. 24 healthy obese participants within three obese class groups; BMI 30-34.9 kg/m2 (n=8), BMI 35-39.9 kg/m2 (n=8), and BMI ≥ 40 kg/m2 (n=8)
2. Male or female adults age 18 to 50 years
3. Weight ≥ 80 kg
4. Estimated creatinine clearance of 60 mL/min to 119 mL/min (n=12) or ≥ 120 mL/min (n=12) (based on the Cockcroft-Gault equation and dosing weight)

Exclusion Criteria:

1. Pregnant or lactating females
2. Significant clinical illness within 3 weeks prior to screening
3. History of severe allergic diseases including drug allergies, with the exception of seasonal allergies
4. Patients initiated on GLP1 agonists
5. Any other factor, condition, or disease, including but not limited to cardiovascular, renal, hepatic, or gastrointestinal disorders that may, in the opinion of the Investigator, jeopardize the safety of the participant or impact the validity of the study results.
6. History of drug addiction or alcohol abuse within the past 12 months
7. Any clinically significant abnormal lab values (Chemistry and Complete Blood Count) during screening
8. Participants unwilling or unable to receive vancomycin by intravenous infusion
9. Individuals with a history of psychiatric or neurological illness, including seizure disorders
10. Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg
11. Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg
12. Pulse rate <50 beats/minute or >100 beats/minute.
13. History of hypersensitivity or infusion reaction to vancomycin, cetirizine, or famotidine
14. Participants with underlying hearing loss
15. Participants that are taking ototoxic drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Probability of target attainment | 24 hours
  Number of participants with a vancomycin area under the concentration-time curve that is between 400 h*mg/L and 600 h*mg/L after a single dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Clinical Research Unit, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pai MP. Antimicrobial Dosing in Specific Populations and Novel Clinical Methodologies: Kidney Function. Clin Pharmacol Ther. 2021 Apr;109(4):952-957. doi: 10.1002/cpt.2179. Epub 2021 Mar 3. PMID 33523498
- [Background] Pai MP. Antimicrobial Dosing in Specific Populations and Novel Clinical Methodologies: Obesity. Clin Pharmacol Ther. 2021 Apr;109(4):942-951. doi: 10.1002/cpt.2181. Epub 2021 Feb 28. PMID 33523485
- [Background] Pai MP, Derstine BA, Lichty M, Ross BE, Sullivan JA, Su GL, Wang SC. Relationships of Vancomycin Pharmacokinetics to Body Size and Composition Using a Novel Pharmacomorphomic Approach Based on Medical Imaging. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e01402-17. doi: 10.1128/AAC.01402-17. Print 2017 Nov. PMID 28807918
- [Background] Crass RL, Dunn R, Hong J, Krop LC, Pai MP. Dosing vancomycin in the super obese: less is more. J Antimicrob Chemother. 2018 Nov 1;73(11):3081-3086. doi: 10.1093/jac/dky310. PMID 30203073
- [Background] Rybak MJ, Le J, Lodise TP, Levine DP, Bradley JS, Liu C, Mueller BA, Pai MP, Wong-Beringer A, Rotschafer JC, Rodvold KA, Maples HD, Lomaestro BM. Therapeutic monitoring of vancomycin for serious methicillin-resistant Staphylococcus aureus infections: A revised consensus guideline and review by the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, the Pediatric Infectious Diseases Society, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2020 May 19;77(11):835-864. doi: 10.1093/ajhp/zxaa036. No abstract available. PMID 32191793